CLINICAL TRIAL: NCT06703632
Title: Evaluation of PreveCol's Efficiency As a Second Line Method for the Early Colorectal Cancer Detection
Acronym: MS-Prevecol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ADVANCED MARKER DISCOVERY S.L. (Industry)
Collaborators: Hospital Universitario Ramon y Cajal (Other); Hospital de Santa Maria, Lisbon (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AMD-CCR-2024-02; 2024-NDMH-5101_240046 (Other Grant/Funding Number: EIT-Health)
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-11

CONDITIONS: Screening for Colon Cancer; Blood Samples; Survey and Questionnaire; Colorectal Carcinoma; Colon Adenocarcinoma; Precancerous Lesion of Colon
Keywords: colorectal cancer; screening programme; liquid biopsy; second line; questionnaire
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Low-risk interventional study
Masking Description: Laboratory Technicians
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PreveCol test after a FOBT positive result (Other): Average-risk participants from the colorectal cancer screening programme with FOBT positive result who are eligible to undergo colonoscopy
  Interventions: Diagnostic Test: blood sampling; Other: Survey using a questionnaire.

INTERVENTIONS:
Diagnostic Test: blood sampling — PreveCol test based on blood sampling
  Other Names: PreveCol
Other: Survey using a questionnaire. — Preference questionnaire for colorectal cancer screening methods
Other: Survey using a questionnaire. — PREMs for colorectal cancer screening programme

SUMMARY:
The objective of this low-risk interventional study is to evaluate whether the PreveCol® test has sufficient efficiency to be considered as a second-line method for the detection of both colorectal cancer and advanced adenomas when used prospectively in the screening population with a previous positive FOBT result, which could include any of the following: both sexes, age 50-69 years, asympthomatic volunteers. The main aims to be answered are:

* Values of efficacy, efficiency, impact and safety of PreveCol.
* Values of preferences of participants for screening methods.
* Values of PREMs into screening programme.

Participants will provide a blood sample prior to a screening colonoscopy, and complete two questionnaires. They will give their sample, information and clinical data to the investigator or health care personnel.

ELIGIBILITY:
Inclusion Criteria:

* Participants ages from 50 to 69 years (both included) at the time of informed consent signed.
* Participants should sign an informed consent. They must understand the nature, significance, implications, and risks of the clinical study before signing the informed consent form.
* Participants with a positive result of FIT/FOBT analysis referred to the gastroenterology department who are eligible to undertake colonoscopy as a regular procedure of the colorectal cancer screening programme.
* Participants asymptomatic, average risk for CRC. Average risk is defined as those individuals who are age 50 or over with no history of adenoma, colorectal cancer, or inflammatory bowel disease, and with no family history of CRC (first degree relatives).

Exclusion Criteria:

* Participants who have developed any another type of cancer in the 5 years prior to their participation in the study.
* Participants who have previously received chemotherapy or radiotherapy (5 years).
* Participants previously or currently diagnosed with Familiar Adenomatous Polyposis or Lynch Syndrome or Inflammatory Bowel Disease.
* Inadequate intestinal preparation for colonoscopy with BBPS score ≤1 in any colon section, excluding diagnostic of CRC.
* Participants who have undergone polypectomy in the previous 5 years.
* Hemolysis of blood sample or absence of blood sample.
* Participants who are arrested at judicial or official request
* Participants who are in a dependent personal or non-medical relationship with the Sponsor or the investigator.

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4538 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | 12 months
  Value of efficiency through the clinical performance (sensitivity, specificity, positive predictive value and negative predictive value) of PreveCol® after FOBT positive result for detecting neoplastic lesions.

SECONDARY OUTCOMES:
Diagnostic performance of cancer | 12 months
  Value of PreveCol's efficiency in second line for detecting cancer
Diagnostic performance of lesions | 12 months
  Value of PreveCol's efficiency in second line for advanced lesions
Value of questionnaires into screening programme | 12 months
  The percentage of number of answers from each preference questions and PREMs

OTHER OUTCOMES:
Safety | 12 months
  Measure the percentage of adverse events and complications directly/indirectly related to interventions of study.

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Albillos, MD, Principal Investigator — Hospital Universitario Ramon y Cajal; Ana Rita, MD, Principal Investigator — Hospital de Santa Maria
Locations (2):
- Hospital de Santa Maria, Lisbon, Lisbon District, Portugal
- Hospital Universitario Ramon y Cajal, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Wagle NS, Cercek A, Smith RA, Jemal A. Colorectal cancer statistics, 2023. CA Cancer J Clin. 2023 May-Jun;73(3):233-254. doi: 10.3322/caac.21772. Epub 2023 Mar 1. PMID 36856579
- [Background] Lordick F, Carneiro F, Cascinu S, Fleitas T, Haustermans K, Piessen G, Vogel A, Smyth EC; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Gastric cancer: ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. Ann Oncol. 2022 Oct;33(10):1005-1020. doi: 10.1016/j.annonc.2022.07.004. Epub 2022 Jul 29. No abstract available. PMID 35914639
- [Background] Greuter MJE, de Klerk CM, Meijer GA, Dekker E, Coupe VMH. Screening for Colorectal Cancer With Fecal Immunochemical Testing With and Without Postpolypectomy Surveillance Colonoscopy: A Cost-Effectiveness Analysis. Ann Intern Med. 2017 Oct 17;167(8):544-554. doi: 10.7326/M16-2891. Epub 2017 Oct 3. PMID 28973514
- [Background] Bujanda L, Sarasqueta C, Castells A, Pellise M, Cubiella J, Gil I, Cosme A, Arana-Arri E, Mar I, Idigoras I, Portillo I; EUSCOLON Study Investigators. Colorectal cancer in a second round after a negative faecal immunochemical test. Eur J Gastroenterol Hepatol. 2015 Jul;27(7):813-8. doi: 10.1097/MEG.0000000000000366. PMID 25856688